CLINICAL TRIAL: NCT02391064
Title: Validation of Brief Computerized Cognitive Assessment in Multiple Sclerosis (BCCAMS) - BICAFMS Study (Brief Cognitive Assessment in French MS Patients)
Brief Title: Validation of Brief Computerized Cognitive Assessment in Multiple Sclerosis (BCCAMS)
Acronym: BICAFMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2013/23
Record Dates: First submitted 2015-02-18; First posted 2015-03-18 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Multiple Sclerosis
Keywords: cognition; brief computerized cognitive assessment; impairment prediction
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient (Experimental): MS Relapsing-remitting under interferon beta-1b treatment in inclusion, Secondary progressive and Primary progressive MS forms
  Interventions: Behavioral: Cognitive evaluation; Behavioral: Expanded Disability Status Scale (EDSS) score
- Control (Experimental): healthy subject
  Interventions: Behavioral: Cognitive evaluation

INTERVENTIONS:
Behavioral: Cognitive evaluation — * Questionnaires for assessment of confounding factors
  * Cognitive evaluation
  * Walking tests and 9 Hole Peg Test
Behavioral: Expanded Disability Status Scale (EDSS) score — - EDSS score
  Arms: Patient

SUMMARY:
Cognitive disorders are common in early stage of Multiple Sclerosis (MS) and concern mainly information processing speed (IPS) which also influences with other cognitive functions such as attention, working memory and executive functions. The investigators validated a computerized test of IPS, the computerized speed cognitive test (CSCT), which can detect disorders of IPS in MS. A short battery was proposed, the brief cognitive assessment for multiple sclerosis (BICAMS) battery, which combines the Symbol-Digit Modalities-test (SDMT), a test of the IPS, and two measures of episodic memory. On the same principle, the investigators propose to validate a short computerized battery to improve the feasibility (brief computerized cognitive assessment (BCCAMS)) combining the CSCT and a computerized test of visual episodic memory.

Purpose: to establish the screening value of a brief computerized cognitive assessment (BCCAMS) combining the computerized speed cognitive test (CSCT) and a new computerized episodic visual memory test (CEVMT) in French-speaking patients with multiple sclerosis as compared to a reference battery (MACFIMS).

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Aged 18-64 years
* Francophone
* MS Relapsing-remitting under interferon beta-1b treatment in inclusion, Secondary progressive and Primary progressive MS forms
* Having signed an informed consent (later than the day of inclusion and before any examination required by research)
* Being affiliated to health insurance

Controls:

* Aged 18-64 years
* Francophone
* Having signed an informed consent (later than the day of inclusion and before any examination required by research)
* Being affiliated to health insurance

Exclusion Criteria:

Patients:

* Other neurological diseases with impact on cognitive functions.
* Severe psychiatric disease or severe depression.
* Current Dependence on alcohol or drugs.
* Modification or stop of psychotropic treatment in less than a month.
* Modification of MS treatment in less than a month.
* Visual, visual-motor and / or motor impairments excluding the ability to perform cognitive tests.
* Pregnant

Controls:

* Neurologic disease and known chronic systemic with impact on cognitive functions.
* Severe psychiatric disease or severe depression.
* Current Dependence on alcohol or drugs.
* Psychotropic treatment
* Cognitive complaint
* Prior cognitive testing with the same tests less than one year.
* Pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 421 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2018-02-18 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
Prediction by the z score BCCAMS of cognitive impairment (at least two tests MACFIMS battery <1.5 SD of control subjects | At the inclusion (Day 0)
  average z scores of CEVMT and CSCT

SECONDARY OUTCOMES:
Determine values of neuropsychological tests in healthy according to age subjects, gender and the level education | At the inclusion (Day 0) and at 1 and 6 months after the inclusion (Day 0)
  BCCAMS and MACFIMS
Ability of the CEVMT to detect episodic memory deficiencies in patients with multiple sclerosis, as compared to established tests of episodic memory | At the inclusion (Day 0) and at 1 and 6 months after the inclusion (Day 0)
  California verbal learning test-II and brief-visual memory test-revised
Correlation between alternate forms of the CEVMT and the Brief visual memory test-revised (BVMT-R) | At the inclusion (Day 0) and at 1 and 6 months after the inclusion (Day 0)
  congnitive test
Prediction between cognitive impairment and occupational status/leisure activities | At the inclusion (Day 0) and 6 months after the inclusion (Day 0)
  questionnaire
Effect of possible confounders on results of cognitive testing, including depression, mood, anxiety and fatigue | At the inclusion (Day 0) and at 1 and 6 months after the inclusion (Day 0)
  scale
Reproducibility of CSCT, CEVMT and the symbol-digit modalities test in clinical settings in patients with multiple sclerosis | At 1 and 6 months after the inclusion (Day 0)
  congnitive test

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital du Bocage, Dijon
  - CH de Dunkerque, Dunkirk
  - Centre Hospitalier Saint Vincent de Paul, Lille
  - Hôpital Roger Salengro, Lille
  - CHU de Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nice, Nice
  - Hôpital Tenon, Paris
  - Hôpital de Poissy Saint Germain, Poissy
  - CHU de Reims, Reims
  - CHU de Strasbourg, Strasbourg